CLINICAL TRIAL: NCT07326085
Title: Pilot Study of MiDialisis App Usage (Estudio Piloto de Uso de MiDiálisis App)
Brief Title: Pilot Study to Evaluate the Feasibility, Adherence and Acceptance of the MiDiálisis Platform for Patients on PD
Acronym: PUMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aida Frías González (Other)
Collaborators: Spanish Society of Nephrology (Other); SOMANE (MADRID SOCIETY OF NEPHROLOGY) (Unknown); Foundation for Biomedical Research of the Hospital Universitario 12 de Octubre (Unknown)
Responsible Party: Sponsor-Investigator, Aida Frías González, M.D., Nephrologist at Universitary Hospital 12 de Octubre, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23/187
Record Dates: First submitted 2025-12-01; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Peritoneal Dialysis (PD)
Keywords: peritoneal dialysys; remote monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INTERVENTION (Experimental): This group will recived the smart band, smart scale and the APP
  Interventions: Device: Smart band; Device: Smart scale; Device: MiDialisis App; Device: Patients will install the app during the phase 2.; Device: Patients will connect the digital scale.; Device: Patients will connect the smartband.

INTERVENTIONS:
Device: Smart band — During Phase 2, patients will use the smart band continuously throughout the day.
Device: Smart scale — During Phase 2, patients will weigh themselves daily using the scale.
Device: MiDialisis App — Patients will enter daily blood pressure data and information related to their peritoneal dialysis therapy.
Device: Patients will install the app during the phase 2. — Patients will download and begin using the application.
Device: Patients will connect the digital scale. — Patients will connect the digital scale to the application via Bluetooth.
Device: Patients will connect the smartband. — Patients will connect the smartband to the application via Bluetooth.

SUMMARY:
The main goal of this study is to assess whether a mobile phone app called MiDiálisis is practical, easy to use, and well-accepted. The app was developed by the Technical University of Madrid (UPM) and is designed to bring together the clinical data of people with chronic kidney disease who are on peritoneal dialysis. This way, both patients and doctors can access the information at any time.

DETAILED DESCRIPTION:
This is a free smartphone app that collects information in three ways:

1. The patient will enter their blood pressure and ultrafiltration values.
2. They will receive a digital scale that sends their weight and body composition to the MiDiálisis app via Bluetooth.
3. They will receive a smartband that sends information about their heart rate, sleep pattern, and physical activity to the MiDiálisis app via Bluetooth.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients with chronic kidney disease who have been on PD for at least 3 months in the same hospital.
* Patients with a stable clinical condition during the 3 months prior to entering the study, defined as no unscheduled hospitalizations or major cardiovascular events (myocardial infarction or stroke) during that period.
* Availability of a smartphone or tablet and internet access for the patient/caregiver.
* Patients who understand the nature of the study and sign the informed consent form.

Exclusion Criteria:

* Patients with limitations for multifrequency body composition measurement (pacemaker or implantable cardioverter defibrillator wearers, and pregnant women).
* Patients who do not routinely use a smartphone or are unfamiliar with the use of mobile applications.
* Patients who are scheduled for a living kidney transplant in the next 6 months.
* Patients with a life expectancy of less than 6 months.
* Patients in a peritoneal ultrafiltration program due to cardiorenal syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-07-27 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility and adherence | The investigators analized the number of times that patient or caregiver access the MiDialisis app during 8 weeks that the patient would be installed the App in his mobile.
  To assess the feasibility and adherence to the use of MiDiálisis among patients undergoing peritoneal dialysis (PD), defined as the number of times per week that the patient or caregiver accesses the MiDiálisis app.

SECONDARY OUTCOMES:
Perceived quality | After 8 weeks of using mobile App (week +16 from recruitment), the patient or caregiver will filled Mobile App Rating Scale (MARS) to analized satisfaction grade.
  To assess patient and caregiver satisfaction (perceived quality, visit 4) with the use of MiDiálisis, measured using the Mobile App Rating Scale (MARS), (23 items, max. 115 points, higher scores mean a better outcome).
Usability | After 8 weeks using MiDialisis dashboard (week +16 from recruitment, visit 4).
  To assess healthcare professionals' satisfaction with the use of the MiDiálisis dashboard. the healthcare professional will filled the System Usability Scale (SUS) (10 items, max 50 points, higher scores mean a better outcome).
In-person Clinical care | At the end of the study (week +24 from recruitment, visit 5).
  Changes in in-person clinical care, measured as the number of face-to-face visits across Phase 1, Phase 2, and Phase 3.
telephone-based clinical care | At the end of the study (week +24 from recruitment, visit 5).
  Changes in telephone-based clinical care, measured as differences in the number of telephone calls across Phase 1, Phase 2, and Phase 3.
unscheduled visits | At the end of the study (week +24 from recruitment, visit 5).
  Changes in the number of unscheduled visits.Measured as the number of unscheduled visits between Phase 1, Phase 2, and Phase 3.
overall clinical care | At the end of the study (week +24 from recruitment, visit 5).
  Changes in overall clinical care. Measured as the number of interactions in the MiDiálisis chat vs. another objetives.
Kidney Disease Quality of Life-36 | At the end of the study (week +24 from recruitment, visit 5).
  Changes in patient-reported health outcomes (PROMs) with MiDiálisis between Phase 1 and Phase 2.
  Measured using the Kidney Disease Quality of Life-36 (KDQOL-36) scale (36 items, max 100 points, higher scores mean a better outcome.).
Kidney Disease and Quality of Life™ Short Form | At the end of the study (week +24 from recruitment, visit 5).
  Changes in patient-reported health experience (PREMS) with the use of MiDiálisis between Phase 1 and Phase 2.
  Measured with the Kidney Disease and Quality of Life™ Short Form (KDQOLSF) (24 items, quantitative, higher scores mean a better outcome).
Pittsburgh Sleep Quality Index | At the end of the study (week +24 from recruitment, visit 5).
  Assess subjective changes in sleep quality between Phase 1 and Phase 2. Measured using the Pittsburgh Sleep Quality Index (PSQI) (19 items, max 21 points, higher scores mean a worse outcome).
Physical Activity Questionnaire | At the end of the study (week +24 from recruitment, visit 5).
  Assess changes in physical activity between Phase 1 and Phase 2. Measured using the International Physical Activity Questionnaire (IPAQ) (7 items, quantitative, higher scores indicate higher levels of physical activity).

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Yuste Lozano, PhD, Principal Investigator — Hospital 12 de Octubre
Locations (1):
- Hospital 12 de Octubre, Madrid, Madrid, Spain